CLINICAL TRIAL: NCT01737632
Title: Family-Based Versus Adolescent Residential Drug Treatment
Brief Title: Family-based and Adolescent Residential Drug Treatment
Acronym: ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Howard Liddle, Professor, University of Miami
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: P50DA011328 (NIH)
Record Dates: First submitted 2012-11-20; First posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Substance Use; Delinquency
Keywords: Adolescents; Residential Treatment; Outpatient Treatment; Substance Abuse; Delinquency; Family Therapy; Multidimensional Family therapy
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multidimensional Family Therapy (MDFT) (Experimental): MDFT is an intensive, in-home family-based drug abuse treatment for adolescent substance abusers. MDFT views family factors in their context -in terms of the network (individual, familial, peer, community) or multiplicity of influences on drug use and change.
  Interventions: Behavioral: Multidimensional Family Therapy (MDFT)
- Adolescent Residential Treatment (Other): The Adolescent Treatment Program (ATP) is a residential dual diagnosed substance abuse treatment program that is staff secure. It is based on a social learning approach which emphasizes positive reinforcement for appropriate coping behavior and social skills, and incorporates a "levels" system which allocates privileges and responsibilities according to the individual's behavioral capacities.
  Interventions: Behavioral: Adolescent Residential Treatment

INTERVENTIONS:
Behavioral: Multidimensional Family Therapy (MDFT) — MDFT assesses and intervenes in five domains: 1) Interventions with the adolescent, 2) interventions with the parent, 3) interventions to improve the parent-adolescent relationship, 4) interventions with other family members, and 5) interventions with external systems.
  Arms: Multidimensional Family Therapy (MDFT)
Behavioral: Adolescent Residential Treatment — The Adolescent Treatment Program targets the adolescent's abuse or dependency on chemicals while simultaneously treating the comorbid symptomatology found in dual diagnosed patients. These goals are accomplished by using four primary forms of intervention: (1) Chemical Education; (2) Group, Individual and Family Counseling; (3) Twelve Step Work; and 4) Psychotropic Medication for Clinical Symptomatology Comorbid with Substance Abuse.
  Arms: Adolescent Residential Treatment

SUMMARY:
The fundamental objective of this study is to compare the effectiveness of an intensive in-home family-based treatment, Multidimensional Family Therapy, with a multifaceted residential treatment, Adolescent Residential Treatment, over 4 years post-intake and to delineate the mechanisms of change for each treatment. The study targets dually- diagnosed adolescent drug abusers recommended for residential treatment.

DETAILED DESCRIPTION:
Aim 1: To compare the effectiveness of residential treatment with outpatient, family-based treatment multiple outcomes including substance use, mental health, school functioning, family function and delinquency among dually diagnosed adolescents.

Hypothesis 1. From intake to 2 months, residential treatment will show better outcomes than the family based treatment. Between 2 months and 18 months, family based treatment will show better outcomes than residential. Between 18 months and four years post intake, outpatient family based treatment will maintain its treatment gains, while the residential treatment condition will show an increase in these same symptoms and behaviors.

Aim 2: To examine the relationship between predictors (family, peer, educational/vocational functioning and involvement in post-treatment services), and outcomes (drug use, co-morbid symptoms, and criminal behavior) during the four-year post intake period.

Hypothesis 2a. Family functioning, educational/vocational functioning, and peer relationships measured at discharge will predict drug use, co-morbid symptoms, and criminal behaviors though the four year longer term follow up period.

Hypothesis 2b. Family functioning, educational/vocational functioning, peer relationships, and involvement in post-treatment services during the post treatment period will predict drug use, co-morbid symptoms, and criminal behavior through the longer term follow up period.

Research Question 1. Is the rate of change in family functioning, educational/vocational functioning, peer relationships, and involvement in post-treatment services related to the rate of change in drug use, co-morbid symptoms, and criminal behavior?

ELIGIBILITY:
Inclusion Criteria:

* Youth between the ages of 13 and 17
* Referred to ATP for residential substance abuse treatment in youth dual diagnosis program
* Dually diagnosed for substance abuse or dependence and at least one of the following co-morbid conditions: major depressive disorder, bipolar disorder, I conduct disorder, oppositional defiant disorder,
* At least one parent or parent-figure can be located at the time of referral.
* Obtain informed consent from a parent or formal guardian and assent from youth to participate in the study.

Exclusion Criteria:

* Have any of the following disorders: Mental Retardation, Eating Disorders, Schizophrenia, or Pervasive Developmental Disorders.
* Current suicidality.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2000-08; Primary Completion 2008-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change in Personal Involvement with Chemicals | Baseline, 2, 4, 12, 18, 24, 36 and 48 months after baseline
  Scale from the Personal Experience Inventory (PEI) developed by Ken Winter.
Change in substance use consumption | Baseline, 2, 4, 12,18,24,36,48 months after intake
  Measure of substance use consumption as measured by the Timeline Follow-back Method.
Change in externalizing symptoms | Baseline, 2, 4, 12, 18, 24, 36 and 48 months
  Externalizing symptoms measured by the Youth Self Report
Change in delinquency | Intake, 2, 4, 12, 18, 24, 35, 48 months after intake
  Measured by youth report on the Self Report Delinquency Scale.
Change in internalzing symptoms | Intake, 2, 4, 12, 18, 24, 36, 48 months after baseline
  Measured by the Youth Self Report (YSR)

SECONDARY OUTCOMES:
Change in family conflict | Baseline, 2, 4, 12, 18, 24, 36, 48 months after baseline
  Parent and youth report on their family conflict as measured by the Family Environment Scale.
Change in parenting practices | Baseline, 2, 4, 12, 18, 24,36, 48 months after baseline
  Measures the extent to which parents monitor, set limits, and provide affection to their teens.
Change in family cohesion | Intake, 2, 4, 12, 18, 24, 26, 48 months after intake
  Youth and parent reports of family closeness measured by the Family Environment Scale (FES)

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Liddle, EdD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami Miller School of Medicine, Miami, Florida
  - The Village, Inc., Miami, Florida

REFERENCES:
- [Background] Zavala SK, French MT, Henderson CE, Alberga L, Rowe C, Liddle HA. Guidelines and challenges for estimating the economic costs and benefits of adolescent substance abuse treatments. J Subst Abuse Treat. 2005 Oct;29(3):191-205. doi: 10.1016/j.jsat.2005.06.004. PMID 16183468